CLINICAL TRIAL: NCT00449384
Title: Severe Impairment Study - Norwegian Version. A Validation and Reliability Study.
Brief Title: SIB-Norwegian Version, Validation and Reliability Study
Status: Completed | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Other Study IDs: F06002
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2007-07

CONDITIONS: Dementia; Diagnostic Tests, Routine
Keywords: Severe Impairment Battery; Clinical Dementia Rating
MeSH Terms: conditions — Dementia | interventions — Diagnostic Screening Programs

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Diagnostic Screening

SUMMARY:
The purpose of this study is to validate and to test interrater reliability for the Norwgian version of Severe Impairment Battery (SIB).

DETAILED DESCRIPTION:
The study will include 60 persons with mild to severe dementia. To test the validation of SIB, we will interview the included persons with Severe Impairment Battery (SIB) and compare the results with Clinical Dementia Rating (CDV)reported by their nurses. To test interrater reliability 30 of the included persons will be interviewed with SIB by two different raters, and the two raters results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Dementia, mild to severe.
* Nursing Home resident

Exclusion Criteria:

* No ability to write or read.
* Physical handicapped, unable to use hands.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-02; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Knut Engedal, PhD, Study Chair — The Norwegian Centre for Dementia Research (NCDR), Norway
Locations (1):
- Sykehuset Innlandet HF - Sanderud, Ottestad, Oppland, Norway